CLINICAL TRIAL: NCT05846763
Title: Efficacy and Safety of Obinutuzumab in Combination With Lenalidomide in Patients With Relapsed and Refractory Follicular Lymphoma (R/R FL): A Prospective Observational Study
Brief Title: Obinutuzumab in Combination With Lenalidomide in Relapsed or Refractory Follicular Lymphoma in Real World Study
Status: Recruiting | Type: Observational
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Other Study IDs: BDHFL2023
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-04

CONDITIONS: Follicular Lymphoma
Keywords: follicular lymphoma; Obinutuzumab; Lenalidomide; real-world
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is planned to prospectively observe and verify the efficacy and safety of induction therapy with obinutuzumab in combination with lenalidomide followed by maintenance therapy with obinutuzumab and lenalidomide in patients with R/R FL in a real-world setting in a Chinese population.

DETAILED DESCRIPTION:
Available data have shown that the combination of obinutuzumab and lenalidomide has shown good efficacy and safety in patients with R/R FL, but the efficacy and safety in Chinese patients remain to be verified.

This study is planned to prospectively observe and verify the efficacy and safety of induction therapy with obinutuzumab in combination with lenalidomide followed by maintenance therapy with obinutuzumab and lenalidomide in patients with R/R FL in a real-world setting in a Chinese population.

The main questions it aims to answer are:

* To assess the ORR in the R/R FL patient population treated with the combination of obinutuzumab and lenalidomide
* To assess CRR, PFS, EFS, DOR, OS, and safety in patients with R/R FL treated with the combination of obinutuzumab and lenalidomide

Participants in this study will not and should not result in any intervention to the patient's treatment and visits. All treatments and visits for patients will be at the physician's discretion according to clinical practice

ELIGIBILITY:
Patients must meet the following criteria for study entry::

* Signed Informed Consent Form
* Age ≥ 18 years at enrollment
* At least one prior line of systemic (Stage III-IV) follicular lymphoma therapy
* Relapsed or refractory to front-line anti-lymphoma therapy; refractory is defined as: tumor shrinkage of less than 50% or disease progression after 4 cycles of standard regimen chemotherapy; response to standard regimen chemotherapy, relapse within 24 months; 2 or more relapses, meeting one of the above criteria as refractory lymphoma.
* Conditional treatment with obinutuzumab in combination with lenalidomide

Exclusion Criteria:

* Patients currently participating or planning to participate in any interventional clinical trial
* Any other reason that, in the opinion of the investigator, makes the patient unsuitable for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include the population of patients with relapsed and refractory follicular lymphoma who are planned to receive the combination of obinutuzumab and Lenalidomide in 9 centers (including 8 sub-centers outside of the Institute of Hematology & Blood Diseases Hospital )
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
overall response rate（ORR） | 24 weeks
  Proportion of patients with complete response (CR) and partial response (PR) after the end of induction therapy.

SECONDARY OUTCOMES:
2-year Progression free survival（PFS24） | Up to 4.5 years
  Time to first disease progression or death from any cause within two years from enrollment.
2-year Event-free survival（EFS24） | Up to 4.5 years
  Time to any event, including disease progression, discontinuation of treatment for any reason, or death within two years from enrollment.
Complete response (CR) | 2.5 years
  Proportion of patients with complete response at the end of treatment
Duration of response (DoR) | Up to 4.5 years
  Time from enrollment to disease progression or death for patients with a complete or partial response
Overall survival (OS) | Up to 4.5 years
  Time to death from any cause from the date of enrollment
Safety(Proportion of Grade 3-4 Hematologic and Non-Hematologic Toxicities) | 4.5 years
  All hematological and non-hematological toxicities from enrollment to 28 days after the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shuhua Yi, Dr, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, Chinese
Locations (1):
- Institute of Hematology and Blood Diseases Hospital ,Chinese Academy of Medical Sciences, Tianjin, China